CLINICAL TRIAL: NCT01327001
Title: Utilization of Fixed Combination (Budesonide/Formoterol and Salmeterol/Fluticasone and Beclomethasone/Formoterol) in Treatment of Asthma Patients in Real Life Condition in Czech Republic (UFO)
Brief Title: Utilization of Fixed Combination (Budesonide/Formoterol and Salmeterol/Fluticasone and Beclomethasone/Formoterol) in Treatment of Asthma Patients
Acronym: UFO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-RCZ-SYM-2010/1
Record Dates: First submitted 2011-03-28; First posted 2011-03-31 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Asthma
Keywords: Asthma bronchiale, fixed combination
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Moderate and severe asthma bronchiale is treated by fixed combination (budesonide/formoterol or salmeterol/fluticasone) in the Czech Republic.

There is a hypothesis that doctors should prescribe to each patients per year: six units of fixed combination budesonide/formoterol, or seven units of fixed combination budesonide/formoterol in approach SMART, or twelve units of fixed combination salmeterol/fluticasone. With regard to current prices the treatment by fixed combination budesonide/formoterol should cost less.

The investigators do not have any data about real life utilization of fixed combination in asthma treatment in Czech Republic The investigators propose to conduct a non-interventional multicentric retrospective epidemiological study looking into the patients records kept by specialist - allergists and pulmologists.

Retrospective data for eligible patients will be reviewed by participating investigators, physicians taking care of their patients, and recorded in the electronic CRF. Only patients who have been treated for asthma bronchiale (classification of severity - moderate or severe persistent asthma) with fixed combination for at least one year could be included into the study. There are no scheduled visits for any patient participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 6 years or over
* Asthma bronchiale, classification of severity - moderate or severe persistent
* Documented fixed combination (budesonide/formoterol or salmeterol/fluticasone) therapy for at least 18 months

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic (specialists in allergology and pulmology)
Sampling Method: Probability Sample
Enrollment: 2815 (Actual)
Dates: Start 2011-04; Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of packs of fixed combination prescribed to patients with asthma bronchiale in one year | 1 year

SECONDARY OUTCOMES:
Asthma severity in patients treated with fixed combination | 1 year
Strength/dose of prescribed fixed combination | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kasak, MD, Principal Investigator — LERYMED spol. s.r.o.
Locations (100):
- Czechia (100):
  - Research Site, Benešov
  - Research Site, Beroun
  - Research Site, Bílovec
  - Research Site, Blansko
  - Research Site, Blovice
  - Research Site, Bohumín
  - Research Site, Brandys N/L
  - Research Site, Brno
  - Research Site, Cheb
  - Research Site, Chomutov
  - Research Site, Chotěboř
  - Research Site, Chrudim
  - Research Site, Čáslav
  - Research Site, Česká Lípa
  - Research Site, České Budějovice
  - Research Site, Český Krumlov
  - Research Site, Český Těšín
  - Research Site, Děčín
  - Research Site, Domažlice
  - Research Site, Fifejdy Ostrava
  - Research Site, Fryštát
  - Research Site, Frýdek-Místek
  - Research Site, Havířov
  - Research Site, Havlíčkův Brod
  - Research Site, Holice
  - Research Site, Horažďovice
  - Research Site, Hořovice
  - Research Site, Hradec Králové
  - Research Site, Hranice
  - Research Site, Jablonec N/N
  - Research Site, Jilemnice
  - Research Site, Jindřichův Hradec
  - Research Site, Kadaň
  - Research Site, Karlovy Vary
  - Research Site, Kladno
  - Research Site, Klatovy
  - Research Site, Kolín
  - Research Site, Kralupy N/V
  - Research Site, Krnov
  - Research Site, Kroměříž
  - Research Site, Kutná Hora
  - Research Site, Liberec
  - Research Site, Litoměřice
  - Research Site, Litomyšl
  - Research Site, Litvnov
  - Research Site, Lochovice
  - Research Site, Lovosice
  - Research Site, MarianskeLazne
  - Research Site, Mělník
  - Research Site, Mladá Boleslav
  - Research Site, Mnichovo Hradiště
  - Research Site, Most
  - Research Site, Náchod
  - Research Site, Neratovice
  - Research Site, Nové Město na Moravě
  - Research Site, Nový Jičín
  - Research Site, Olomouc
  - Research Site, Opava
  - Research Site, Orlová
  - Research Site, Ostrava
  - Research Site, Ostrava - Hrabuvka
  - Research Site, Pardubice
  - Research Site, Pelhřimov
  - Research Site, Pilsen
  - Research Site, Písek
  - Research Site, Poděbrady
  - Research Site, Prachatice
  - Research Site, Prague
  - Research Site, Prostejov - Karlov
  - Research Site, Prostějov
  - Research Site, Přerov
  - Research Site, Příbor
  - Research Site, Příbram
  - Research Site, Rakovník
  - Research Site, Roudnice N/L
  - Research Site, Rožnov pod Radhoštěm
  - Research Site, Rychnov nad Kněžnou
  - Research Site, Slaný
  - Research Site, Sokolov
  - Research Site, Stod
  - Research Site, Strakonice
  - Research Site, Svitavy
  - Research Site, Šumperk
  - Research Site, Tachov
  - Research Site, Tábor
  - Research Site, Teplice
  - Research Site, Trutnov
  - Research Site, Třebíč
  - Research Site, Třemošná
  - Research Site, Týn nad Vltavou
  - Research Site, Ústí nad Labem
  - Research Site, Valašské Meziříčí
  - Research Site, Vsetín
  - Research Site, Vyškov
  - Research Site, Zdar
  - Research Site, Zlín
  - Research Site, Znojmo
  - Research Site, Žamberk
  - Research Site, Žatec
  - Research Site, Železný Brod